CLINICAL TRIAL: NCT00660816
Title: Randomized Phase II Trial, Comparing Standard of Care Chemotherapy (Pemetrexed or Docetaxel) Plus Erlotinib to Standard of Care Chemotherapy (Pemetrexed or Docetaxel) Alone in EGFR TKI-Responsive Non-Small Cell Lung Cancer
Brief Title: Pemetrexed or Docetaxel With or Without Erlotinib in Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE2507; P30CA043703 (NIH); CASE2507 (Other: Case Comprehensive Cancer Center); CASE-2507-CC350 (Other: Cancer Center IRB)
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive pemetrexed disodium IV over 10 minutes OR docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients may continue to receive standard chemotherapy with or without erlotinib hydrochloride in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pemetrexed disodium; Drug: docetaxel
- Arm II (Experimental): Patients receive pemetrexed disodium IV over 10 minutes OR docetaxel IV over 60 minutes on day 1 and erlotinib hydrochloride PO once daily on days 2-19. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients may continue to receive standard chemotherapy with or without erlotinib hydrochloride in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: pemetrexed disodium; Drug: docetaxel

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally once daily on days 2-19.
  Other Names: erlotinib
  Arms: Arm II
Drug: pemetrexed disodium — Given IV over 10 minutes on day 1
  Other Names: MTA
Drug: docetaxel — IV over 60 minutes on day 1.
  Other Names: TXT

SUMMARY:
RATIONALE: Pemetrexed disodium and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving pemetrexed disodium or docetaxel together with erlotinib hydrochloride is more effective than giving pemetrexed disodium or docetaxel alone in treating non-small lung cancer.

PURPOSE: This randomized phase II trial is studying how well giving pemetrexed disodium or docetaxel together with or without erlotinib hydrochloride works in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate whether maintenance erlotinib hydrochloride added to standard of care (pemetrexed disodium or docetaxel) chemotherapy in patients with erlotinib hydrochloride-responsive advanced non-small cell lung cancer leads to an improved progression-free survival as compared to standard of care pemetrexed disodium or docetaxel alone.

Secondary

* To evaluate the effect of maintenance erlotinib hydrochloride on the response rate to standard of care (pemetrexed disodium or docetaxel) therapy in patients with erlotinib hydrochloride-responsive advanced non-small cell lung cancer as compared to standard of care (pemetrexed disodium or docetaxel) alone.
* To evaluate whether maintenance erlotinib hydrochloride added to standard of care (pemetrexed disodium or docetaxel) chemotherapy in patients with erlotinib hydrochloride-responsive advanced non-small cell lung cancer leads to an improved overall survival as compared to standard of care (pemetrexed disodium or docetaxel) alone.
* To evaluate the effect of maintenance erlotinib hydrochloride on the disease stabilization (complete response [CR] + partial response [PR] + stable disease [SD]) rate to standard of care (pemetrexed disodium or docetaxel) therapy in patients with erlotinib hydrochloride-responsive advanced non-small cell lung cancer as compared to standard of care (pemetrexed disodium or docetaxel) alone.
* To evaluate the utility of early positron emission tomography (PET) scanning (baseline versus 1 cycle of protocol therapy) on overall disease assessment and prediction of treatment responsiveness.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to lifetime smoking status (never vs ever) and ECOG performance status (0-1 vs ≥ 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: (standard of care alone): Patients receive pemetrexed disodium intravenously (IV) over 10 minutes OR docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: (standard of care plus erlotinib): Patients receive pemetrexed disodium IV over 10 minutes OR docetaxel IV over 60 minutes on day 1 and erlotinib hydrochloride orally (PO) once daily on days 2-19. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients may continue to receive standard chemotherapy with or without erlotinib hydrochloride in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8 weeks.

ELIGIBILITY:
INCLUSION CRITERIA

* Pathologic diagnosis of stage IIIB (with pleural effusion) or IV non-small cell lung cancer
* Progression following at least twelve weeks of treatment with single-agent erlotinib (or in combination with other experimental agents) during which time the patients experienced a clinical benefit as assessed by his/her treating physician and corroborated by radiographic assessment (at least one CT scan following at least 4 weeks of erlotinib monotherapy demonstrating stable disease or response on erlotinib therapy).
* At least one measurable lesion as defined by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy of at least 12 weeks
* Absolute neutrophil count (ANC) >= 1.5x10(9)/L
* Platelet count >= 100x 10(9)
* Hemoglobin >= 8.0 g/dl
* Serum creatinine =< 1.5 upper limit of normal OR calculated creatinine clearance >= 45 mL/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Available baseline diagnostic tumor specimen for correlative studies, any diagnostic material will be acceptable- paraffin block, cell block, fine needle aspirate etc.
* Patients must provide verbal and written informed consent to participate in the study
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Patient must be able to take folic acid, vitamin B12 as well as dexamethasone therapy as per protocol guidelines
* Patient must be able to interrupt nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed (this exclusion criteria applies only to patients who have not received pemetrexed chemotherapy prior)

EXCLUSION CRITERIA

* Active central nervous system disease (CNS) metastases, as indicated by clinical symptoms, cerebral edema or progressive growth (subjects with a clinical history of CNS metastases or cord compression are allowable if they have been definitively treated and are clinically stable for at least 4 weeks before first dose of study treatment for prior whole brain radiation and 2 weeks for prior gamma knife therapy)
* More than 1 prior cytotoxic chemotherapy regimen for relapsed or metastatic disease (not including erlotinib)
* Any prior epidermal growth factor receptor (EGFR) inhibitor therapy except for erlotinib
* Major surgery, chemotherapy, or investigational agents within 3 weeks of treatment day 1 (except for erlotinib). Radiation therapy within 2 weeks of treatment day 1 (except for erlotinib).
* Prior treatment with both pemetrexed and docetaxel chemotherapy
* Pregnancy or breastfeeding or not receiving adequate contraception (including the patients spouse)
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Patients who must receive pemetrexed and have the presence of third space fluid which cannot be controlled by drainage
* Patients who must receive docetaxel and who have peripheral neuropathy > grade 2
* Patients who must receive docetaxel and who have had a hypersensitivity reaction to medications formulated with polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2013-04 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (13):
- United States (13):
  - Wayne State University, Detroit, Michigan
  - Columbia Presbyterian, New York, New York
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - UH-Monarch, Mayfield Heights, Ohio
  - UH-Firelands, Sandusky, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Alimta or Taxotere alone
- Experimental: Alimta or Taxotere and Tarceva
Period: Overall Study
Arm/Group | Active Comparator | Experimental
Started | 24 | 22
Completed | 4 | 3
Not Completed | 20 | 19
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Disease Progression | 16 | 12
Not completed — Complicating Disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Experimental | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Full Range); unit: years] | 67.0 (11.08) [44 to 83] | 63.6 (10.62) [46 to 84] | 65.3 (10.78) [44 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 4 | 5
  White | 20 | 15 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: From the date of randomization to the date of disease progression or the date of death, whichever occurs first and censored at the date of last followed for those survivors without disease progression.
Time Frame: 18 months after enrollment of last patient
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 22
Months | 5.5 [2.6 to 6.6] | 4.4 [2.9 to 7.5]

2. Secondary Outcome: Overall Survival
Description: Measured from the date of randomization to the date of death, whichever occurs first and censored at the date of last followed for those survivors
Time Frame: 36 months after enrollment of last patient
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 22
Months | 16.4 [6.6 to 39] | 14.2 [7 to 23.9]

3. Secondary Outcome: Response Rate
Description: Estimated based on the number of responses by excluding the dropouts who are not evaluable for response using a binomial distribution
Time Frame: 36 months after enrollment of last evaluable patient
Population: Patients with a complete response, partial response, stable disease, or progressive disease
Measure: Number; unit: participants
Arm/Group | Active Comparator | Experimental
Number analyzed (Participants) | 15 | 18
participants | 2 | 3

4. Secondary Outcome: Disease Stabilization Rate (e.g., Complete Response, Partial Response, and Stable Disease)
Description: Estimated based on number of evaluable patients with complete response, partial response or stable disease
Time Frame: 36 months after enrollment of last patient
Population: Patients with a complete response, partial response, stable disease, or progressive disease
Measure: Number; unit: participants
Arm/Group | Active Comparator | Experimental
Number analyzed (Participants) | 15 | 18
participants | 15 | 16

ADVERSE EVENTS:
Arm/Group | Active Comparator | Experimental
Serious Adverse Events (participants affected / at risk) | 4/24 | 17/22
Other Adverse Events (participants affected / at risk) | 24/24 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator (N=24) | Experimental (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Crohn's exacerbation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator (N=24) | Experimental (N=22)
Constipation (Gastrointestinal disorders) | 12 (17) | 8 (13)
Nausea (Gastrointestinal disorders) | 10 (16) | 8 (18)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 11 (17)
Vomiting (Gastrointestinal disorders) | 3 (4) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's exacerbation (Gastrointestinal disorders) | 0 (0) | 1 (5)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (25) | 15 (64)
White blood cell decreased (Investigations) | 10 (37) | 12 (43)
Aspartate aminotransferase increased (Investigations) | 9 (11) | 6 (12)
Neutrophil count decreased (Investigations) | 8 (24) | 7 (21)
Alkaline phosphatase increased (Investigations) | 5 (7) | 7 (8)
Alanine aminotransferase increased (Investigations) | 3 (3) | 7 (9)
Platelet count decreased (Investigations) | 4 (10) | 6 (19)
Weight loss (Investigations) | 1 (1) | 5 (8)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (3) | 2 (2)
Weight gain (Investigations) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (16) | 11 (27)
Anorexia (Metabolism and nutrition disorders) | 8 (14) | 8 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8) | 6 (11)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 4 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 14 (29) | 13 (28)
Edema limbs (General disorders) | 6 (10) | 3 (4)
Non-cardiac chest pain (General disorders) | 5 (5) | 4 (4)
Pain (General disorders) | 2 (3) | 5 (6)
Fever (General disorders) | 3 (3) | 3 (3)
Chills (General disorders) | 2 (2) | 3 (3)
Flu like symptoms (General disorders) | 1 (1) | 1 (1)
Localized edema (General disorders) | 1 (1) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (14) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (11)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Epistaxis (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (4) | 7 (46)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
"Skin and subcutaneous tissue disorders - Other, specify" (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 11 (29) | 11 (23)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
"Musculoskeletal and connective tissue disorder - Other, specify" (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (10) | 7 (13)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 3 (4)
Confusion (Psychiatric disorders) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 2 (2)
Dizziness (Nervous system disorders) | 3 (5) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Lung infection (Infections and infestations) | 2 (2) | 1 (3)
"Infections and infestations - Other, specify" (Infections and infestations) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (3)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 3 (4) | 1 (1)
Hot flashes (Vascular disorders) | 4 (4) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 3 (4) | 2 (2)
Watering eyes (Eye disorders) | 2 (2) | 3 (5)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
"Eye disorders - Other, specify" (Eye disorders) | 0 (0) | 1 (1)
"Renal and urinary disorders - Other, specify" (Renal and urinary disorders) | 2 (2) | 2 (4)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 3 (4)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
"Ear and labyrinth disorders - Other, specify" (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes